CLINICAL TRIAL: NCT04486833
Title: A Phase 1/2 Open-Label, Dose-Escalation and Clinical Response Study of Quaratusugene Ozeplasmid in Combination With Osimertinib in Patients With Advanced, Metastatic EGFR-Mutant, Metastatic Non-Small Cell Lung Cancer
Brief Title: Quaratusugene Ozeplasmid (Reqorsa) and Osimertinib in Patients With Advanced Lung Cancer Who Progressed on Osimertinib
Acronym: Acclaim-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genprex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONC-003
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Non-Small Cell Lung
Keywords: Epidermal growth factor receptor mutation (EGFR); osimertinib; Tumor suppressor gene 2 (TUSC2); Lipid nanoparticle (LNP); Gene therapy; Tagrisso; FUS1-nanoparticles; NSCLC; Reqorsa; quaratusugene ozeplasmid
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Platinum Compounds; Cisplatin; Carboplatin

STUDY DESIGN:
Intervention Model Description: Phase 1: 3+3 dose escalation to identify RP2D.
  Phase 2: RP2D further evaluated in Phase 2a expansion followed by parallel randomization in a 1:1 ratio to either investigational arm or control arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational (Experimental): In Phase 1, Phase 2a and the investigational arm of Phase 2b, patients will receive their assigned dose of quaratusugene ozeplasmid (intravenous administration once every 21 days) plus osimertinib (80 mg fixed dose oral tablet taken daily starting on Day 1 through Day 21 of every 21-day treatment cycle) until disease progression or unacceptable toxicity.
  Interventions: Biological: quaratusugene ozeplasmid; Drug: osimertinib
- Control (Active Comparator): In the control arm of Phase 2b, patients will receive platinum-based chemotherapy until disease progression or unacceptable toxicity.
  Interventions: Drug: Platinum-Based Chemotherapy

INTERVENTIONS:
Biological: quaratusugene ozeplasmid — Quaratusugene ozeplasmid is an experimental non-viral immunogene therapy utilizing the TUSC2 gene, designed to target cancer cells by interrupting cell signaling pathways that allow cancer cells to grow, reestablishing pathways that promote cancer cell death and modulating the immune response against cancer cells.
  Other Names: Reqorsa
  Arms: Investigational
Drug: osimertinib — Osimertinib is a 3rd generation EGFR tyrosine kinase inhibitor (TKI) oral tablet administered daily, as indicated for treatment of patients with metastatic NSCLC whose tumors have EGFR genetic deletions or mutations.
  Other Names: Tagrisso
  Arms: Investigational
Drug: Platinum-Based Chemotherapy — Cisplatin and carboplatin are intravenously administered platinum agents that are combined with other cytotoxic chemotherapy agents such as pemetrexed.
  Other Names: cisplatin; carboplatin
  Arms: Control

SUMMARY:
The purpose of this randomized study is to determine the safety and efficacy of quaratusugene ozeplasmid (Reqorsa) added to osimertinib in NSCLC patients with activating EGFR mutations who have progressed while on treatment with osimertinib. Quaratusugene ozeplasmid consists of non-viral lipid nanoparticles that encapsulate a DNA plasmid with the TUSC2 tumor suppressor gene and is the first systemic gene therapy for cancer.

The study is comprised of a Phase 1 dose escalation portion and two Phase 2 portions evaluating safety and efficacy. Enrollment in the Phase 1 dose escalation portion is complete and the recommended Phase 2 dose (RP2D) was determined. Phase 2a has initiated and enrolled patients are treated with quaratusugene ozeplasmid at the RP2D in combination with osimertinib. In Phase 2b, patients will be randomized to receive either quaratusugene ozeplasmid plus osimertinib or platinum-based chemotherapy.

DETAILED DESCRIPTION:
Acclaim-1 is an open-label, multi-center, Phase 1/2 study evaluating quaratusugene ozeplasmid (Reqorsa) plus osimertinib (investigational arm) versus platinum-based chemotherapy (control arm) in patients with advanced metastatic or recurrent NSCLC.

Toxicities will be assessed by the Investigator using United States National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. Serious Adverse Events and Dose Limiting Toxicities (DLT) will be reviewed by a Safety Review Committee.

Phase 1 - Dose Escalation: The RP2D of quaratusugene ozeplasmid when given in combination with osimertinib has been identified.

Phase 2a: This expansion cohort will be enrolled to better characterize safety, tolerability, and preliminary anti-tumor activity of the combination therapy.

Phase 2b: Quaratusugene ozeplasmid in combination with osimertinib will be further evaluated using the RP2D identified in Phase 1. Patients may receive local therapy, such as radiation therapy, to progressing lesions prior to enrollment. Patients will be randomized to receive either the investigational arm or the control arm in a 1 to 1 ratio and stratified based on prior local radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Histologically or cytologically documented NSCLC.
3. Stage III or IV NSCLC or recurrent NSCLC that is not potentially curable by radiotherapy or surgery.
4. The NSCLC must be epidermal growth factor receptor (EGFR) mutation positive-positive based on results from most recent tissue biopsy or most recent evaluation of circulating tumor DNA.
5. Achieved clinical response to osimertinib for ≥4 months, which can be a response of stable disease. Must have a minimum of a 10-day osimertinib washout completed at the time of enrollment.
6. Must have radiological progression on osimertinib treatment and can have either asymptomatic disease or symptomatic disease. In addition:

   1. Must have measurable disease per RECIST 1.1.
   2. Must have progression on osimertinib treatment as a single agent or in combination with other anti-cancer agents as their most recent treatment.

   Notes:
   * Patients may have had treatment with other EGFR inhibitors as single agents prior to osimertinib.
   * Patients may have progression on osimertinib treatment being used for adjuvant therapy after surgery.
7. Eastern Cooperative Oncology Group performance status (ECOG PS) score from 0 to 1.
8. Must be ≥28 days beyond major surgical procedures such as thoracotomy, laparotomy, or joint replacement and must not have evidence of wound dehiscence, active wound infection, or comparable major residual complications of the surgery per Investigator assessment.
9. Asymptomatic brain metastases must meet ALL criteria of the following (a-d):

   1. No history of seizures in the preceding six months.
   2. Definitive treatment must be completed ≥21 days.
   3. Must be off steroids administered because of brain metastases or related symptoms for ≥7 days.
   4. Post-treatment imaging must demonstrate stability or regression of the brain metastases.
10. Must have and be willing to submit a prior tumor biopsy or undergo a biopsy during Screening to obtain tumor tissue for submission to a central laboratory for IHC analysis and FISH or qPCR testing.
11. Absolute neutrophil count (ANC) >1500/mm3, platelet count >100,000/mm3 within ≤28 days.
12. Adequate renal function documented by serum creatinine of ≤1.5 mg/dL or calculated creatinine clearance >50 ml/min within ≤28 days.
13. Adequate hepatic function as documented by serum bilirubin <1.5 mg/dL and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 X upper limit of normal (ULN) within ≤28 days.
14. Stable cardiac condition with a left ventricular ejection fraction ≥40% within ≤28 days.
15. If female of childbearing potential (FOCBP), must have negative serum pregnancy test (serum beta-human chorionic gonadotropin [β-hCG]) within ≤7 days.
16. FOCBP and non-sterile male patients with female partner(s) of childbearing potential must agree to use two forms of contraception including one highly effective and one effective method beginning ≥2 weeks prior to enrollment through four months following the last dose of study treatment.
17. If male, must agree to no sperm donation during study treatment and for an additional four months following the last dose of study treatment.
18. Must have voluntarily signed an informed consent in accordance with institutional policies.

Exclusion Criteria:

1. Unable to tolerate osimertinib treatment, leading to early treatment discontinuation or prolonged/frequent dosage modifications as determined by the Investigator.
2. Received prior gene therapy.
3. Other genetic characteristics (such as ALK, ROS, BRAF V600E mutations) which make them a candidate for treatment with other approved targeted therapies.
4. Received radiotherapy to the skull, spine, thorax, or pelvis within ≤30 days.
5. Active concurrent malignancies, i.e., cancers other than NSCLC that require systemic therapy.
6. Active systemic viral, bacterial, or fungal infection(s) requiring treatment.
7. Serious concurrent illness or psychological, familial, sociological, geographical, or other concomitant conditions that, in the opinion of the Investigator, would not permit adequate follow-up and compliance with the study protocol.
8. History of myocardial infarction or unstable angina within ≤6 months.
9. Known human immunodeficiency virus (HIV) infection or has active hepatitis infection.
10. Female who is pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2021-09-03 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) - Phase 1 | First 21-day treatment cycle for each dose level cohort
  RP2D, which will be the maximum tolerated dose (MTD) or, if the MTD is not defined by the safety data, RP2D will be determined based on an integrated assessment of all available clinical safety and preliminary efficacy data.
Overall Response Rate (ORR) - Phase 2a | Approximately 3 months
  ORR (complete response [CR]+ partial response [PR]) according to RECIST using best overall response.
Progression-free Survival (PFS) - Phase 2b | Approximately 11 months
  PFS from randomization to disease progression or death. Response according to RECIST.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) - Phase 1 | Approximately 9 months
  PFS from first dose to disease progression or death. Response according to RECIST.
Overall Response Rate (ORR) - Phase 1 | Approximately 3 months
  ORR (CR+ PR) according to RECIST using best overall response.
Duration of Response (DOR) - Phase 1 | Approximately 9 months
  DOR (CR + PR) from response to disease progression. Response according to RECIST.
Pharmacokinetics (PK) of Quaratusugene Ozeplasmid - Phase 1 | First 21-day treatment cycle
  Concentration of quaratusugene ozeplasmid in whole blood samples.
Progression-free Survival (PFS) - Phase 2a | Approximately 11 months
  PFS from first dose to disease progression or death. Response according to RECIST.
Time to Progression (TTP) - Phase 2a | Approximately 11 months
  TTP from first dose to disease progression. Response according to RECIST.
Overall Survival (OS) - Phase 2a | Approximately 21 months
  OS from first dose until death or discontinuation due to withdrawal of consent.
Pharmacokinetics (PK) of Quaratusugene Ozeplasmid - Phase 2a | Approximately 22 days
  Concentration of quaratusugene ozeplasmid in whole blood samples.
Overall Response Rate (ORR) - Phase 2b | Approximately 3 months
  ORR (CR+ PR) according to RECIST using best overall response.
Time to Progression (TTP) - Phase 2b | Approximately 11 months
  TTP from first dose to disease progression. Response according to RECIST.
Duration of Response (DOR) - Phase 2b | Approximately 11 months
  DOR (CR + PR) according to RECIST from response to disease progression.
Overall Survival (OS) - Phase 2b | Approximately 21 months
  OS from randomization to death or discontinuation due to withdrawal of consent.
Incidence of Adverse Events - Phase 2b | Approximately 11 months
  Treatment-related adverse events (AEs) graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events.
Pharmacokinetics (PK) of Quaratusugene Ozeplasmid - Phase 2b | Approximately 22 days
  Concentration of quaratusugene ozeplasmid in whole blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. Berger, MD, Study Director — Genprex, Inc.
Locations (10):
- United States (10):
  - Valkyrie Clinical Trials, Los Angeles, California
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Carle Cancer Institute, Urbana, Illinois
  - Markey Cancer Center, Lexington, Kentucky
  - Maryland Oncology Hematology, Rockville, Maryland
  - The Valley Hospital - Luckow Pavilion, Paramus, New Jersey
  - Gabrail Cancer Center Research, Canton, Ohio
  - Millennium Oncology, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spira AI, Berz D, Jotte RM, Pachipala KK, Berger MS. Dose Escalation Trial of the Combination of Osimertinib and Quaratusugene Ozeplasmid Gene Therapy in Patients with Advanced NSCLC. Clin Lung Cancer. 2025 Nov 17;27(1):75-81. doi: 10.1016/j.cllc.2025.11.009. Online ahead of print. PMID 41385873
- See also: Dose Escalation Trial of the Combination of Osimertinib and Quaratusugene Ozeplasmid Gene Therapy in Patients with Advanced NSCLC — https://www.clinical-lung-cancer.com/article/S1525-7304%2825%2900317-1/fulltext